CLINICAL TRIAL: NCT03020810
Title: Dupilumab Compassionate Use Study
Status: Approved for marketing | Type: Expanded Access
Sponsor: Sally E. Wenzel MD (Other)
Responsible Party: Sponsor-Investigator, Sally E. Wenzel MD, Professor of Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Other Study IDs: PRO16120334
Record Dates: First submitted 2017-01-11; First posted 2017-01-13 (Estimated); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — dupilumab

INTERVENTIONS:
Drug: Dupilumab — The patient will receive a 600 mg subcutaneous dupilumab loading dose on Day 1, and then 300 mg subcutaneous dupilumab every 2 weeks

SUMMARY:
This is a single patient expanded access, compassionate and non-emergency use study that provides patients with severe asthma, who do not qualify for ongoing clinical trials with dupilumab, access to this investigational treatment.

DETAILED DESCRIPTION:
This study is being undertaken to determine whether dupilumab has efficacy in extremely severe asthma, and to allow a very severe asthma patient, who has been tried on nearly every immunosuppressive drug, early access to a potentially effective therapy.

The patient will continue in the study indefinitely. Safety will be evaluated and serious adverse events will be reported.

ELIGIBILITY:
Inclusion Criteria:

* Sever systemic corticosteroid dependent asthma for more than 5 years

Exclusion Criteria:

* Disease other than asthma
* Circulation eosinophils more than 1500/ul
* Current smoker or more than 10 pack years

This is a single-patient study. The University of Pittsburgh site is not enrolling new patients.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult